CLINICAL TRIAL: NCT00005046
Title: A Phase I Open Label Assessment of the Safety and Pharmacokinetics of Intraperitoneal PACLIMER Microspheres (Polilactofate/Paclitaxel) in Patients With Ovarian Cancer
Brief Title: Paclitaxel in Treating Patients With Recurrent or Persistent Ovarian or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: GOG Foundation (Network)
Purpose: Treatment
Other Study IDs: CDR0000067638; GOG-9904; GP-700-9901
Record Dates: First submitted 2000-04-06; First posted 2003-11-04 (Estimated); Last update posted 2013-05-27 (Estimated); Status verified 2008-07

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: recurrent ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial | interventions — Drug Therapy; Paclitaxel

INTERVENTIONS:
Drug: chemotherapy
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase I trial to study the effectiveness of paclitaxel in treating patients who have recurrent or persistent ovarian or primary peritoneal cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the safety and tolerability of intraperitoneal administration of paclitaxel (Paclimer microspheres) in patients with recurrent or persistent ovarian or primary peritoneal carcinoma. II. Determine and confirm the maximum tolerated dose of this regimen in this patient population. III. Determine plasma paclitaxel concentrations at selected times after intraperitoneal administration of Paclimer microspheres in these patients.

OUTLINE: This is a dose escalation study. Patients receive intraperitoneal paclitaxel (Paclimer microspheres) every 8 weeks for 2 courses. Cohorts of 1-3 patients receive escalating doses of intraperitoneal paclitaxel (Paclimer microspheres) until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 patients experience dose limiting toxicities. Once the probable MTD is determined, an additional cohort of 8 patients is accrued to confirm the MTD. The MTD is confirmed as the dose level at which at least 6 of 8 patients demonstrate acceptable safety and tolerability.

PROJECTED ACCRUAL: A maximum of 24 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Recurrent or persistent ovarian and/or primary peritoneal carcinoma Adequate potential intraperitoneal fluid distribution with no gross fluid loculations and adhesions that would significantly affect intraperitoneal drug distribution

PATIENT CHARACTERISTICS: Age: 21 and over Performance status: GOG 0-2 Life expectancy: At least 6 months Hematopoietic: Absolute neutrophil count at least 1,500/mm3 WBC at least 3,000/mm3 Platelet count at least 100,000/mm3 Granulocyte count at least 1,500/mm3 Hepatic: Bilirubin no greater than 1.5 times upper limit of normal Renal: Creatinine less than 2.0 mg/dL Other: No other sufficiently severe medical problems unrelated to malignancy that would preclude study compliance or cause exposure to undue risks No prior unmanageable reaction to paclitaxel

PRIOR CONCURRENT THERAPY: Biologic therapy: Not specified Chemotherapy: At least 4 weeks since prior myelosuppressive chemotherapy (6 weeks for nitrosourea and mitomycin) and recovered Endocrine therapy: Not specified Radiotherapy: At least 4 weeks since prior radiotherapy to major bone marrow containing areas Surgery: Not specified Other: At least 1 month since other prior investigational agents

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-04; Primary Completion 2007-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deborah K. Armstrong, MD, Study Chair — Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins
Locations (5):
- United States (5):
  - Chao Family Comprehensive Cancer Center, Orange, California
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Indiana University Cancer Center, Indianapolis, Indiana
  - Washington University School of Medicine, St Louis, Missouri
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio

REFERENCES:
- [Result] Armstrong DK, Fleming GF, Markman M, Bailey HH. A phase I trial of intraperitoneal sustained-release paclitaxel microspheres (Paclimer) in recurrent ovarian cancer: a Gynecologic Oncology Group study. Gynecol Oncol. 2006 Nov;103(2):391-6. doi: 10.1016/j.ygyno.2006.02.029. Epub 2006 Apr 19. PMID 16626792